CLINICAL TRIAL: NCT02505763
Title: Treatment of Pleural Effusion by Routine Thoracic Ultrasound
Brief Title: Thoracic Ultrasound in the Treatment of Pleural Effusion
Acronym: ECHOPLEV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/14/7418
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strategy with thoracic ultrasound (Experimental): * Use of thoracic ultrasound for the treatment of pleural effusion, treatment and monitoring.
  * Use of other examinations like chest CT if necessary
  Interventions: Procedure: Strategy with thoracic ultrasound
- Strategy without thoracic ultrasound (No Intervention): * Usual care : without thoracic ultrasound
  * Use of chest radiography or chest CT scan if necessary, as for treatment and monitoring.
  Usual care: without the use of ultrasound Using either chest radiography or TDM if necessary, as for treatment and monitoring.

INTERVENTIONS:
Procedure: Strategy with thoracic ultrasound — This strategy involves the systematic use of thoracic ultrasound for the treatment of pleural effusion, treatment and follow up care.
  Arms: Strategy with thoracic ultrasound

SUMMARY:
The main objective of the study is to assess the cost-effectiveness ratio of two management strategies of pleurisy in adults : a strategy by systematic thoracic ultrasound versus a strategy without thoracic ultrasound.

DETAILED DESCRIPTION:
Comparison of two management strategies pleural effusions from diagnosis and during the first year of follow up care.

Patients are randomized into two groups, each group receiving a different management strategy.

Both strategies are compared:

Strategy A that involves the systematic use of thoracic ultrasound for the treatment of pleural effusion, treatment and follow up care. It will be possible to have recourse to other tests (such as chest CT) if deemed necessary by the practitioner.

Strategy B, which consists of the usual care pleurisy and thus without use of ultrasound: gestures are guided either by chest radiograph or by CT chest as necessary in the treatment and monitoring. A systematic radiographic pleural after each gesture is performed.

The management is inspired by the English recommendations currently validated and applied in Anglo-Saxon countries.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized or seen in consultation with pleural effusion diagnosed clinically or radiologically whatever be its initial management.

Exclusion Criteria:

* Patient with a neoplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The cost-effectiveness ration | 1 year
  Cost estimates will be conducted from the perspective of health insurance. The expenses incurred in the care of patients with pleurisy will be counted in both groups during the follow-up year.
  The effectiveness will be assessed against the complications of strategy (pneumothorax, respiratory sequelae, surgery, mortality, chest pain sequelae, radiological consequences).

SECONDARY OUTCOMES:
The duration of hospitalization | 1 year
  number of day of hospitalization between the two strategies

OTHER OUTCOMES:
The irradiation rate | 1 year
  calculation of irradiation rate between the two strategies
Number of consultations | 1 year
  The number of consultations between the two strategies

CONTACTS AND LOCATIONS:
Overall Officials: Elise NOEL-SAVINA, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- NOEL-SAVINA Elise, Toulouse, Midi Pyrenees, France

REFERENCES:
- [Background] Havelock T, Teoh R, Laws D, Gleeson F; BTS Pleural Disease Guideline Group. Pleural procedures and thoracic ultrasound: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii61-76. doi: 10.1136/thx.2010.137026. No abstract available. PMID 20696688
- [Background] Reissig A, Copetti R, Mathis G, Mempel C, Schuler A, Zechner P, Aliberti S, Neumann R, Kroegel C, Hoyer H. Lung ultrasound in the diagnosis and follow-up of community-acquired pneumonia: a prospective, multicenter, diagnostic accuracy study. Chest. 2012 Oct;142(4):965-972. doi: 10.1378/chest.12-0364. PMID 22700780
- [Background] Jones PW, Moyers JP, Rogers JT, Rodriguez RM, Lee YC, Light RW. Ultrasound-guided thoracentesis: is it a safer method? Chest. 2003 Feb;123(2):418-23. doi: 10.1378/chest.123.2.418. PMID 12576360
- [Background] Ikezoe J, Morimoto S, Arisawa J, Takashima S, Kozuka T, Nakahara K. Percutaneous biopsy of thoracic lesions: value of sonography for needle guidance. AJR Am J Roentgenol. 1990 Jun;154(6):1181-5. doi: 10.2214/ajr.154.6.2110724.
- [Background] Chen HJ, Yu YH, Tu CY, Chen CH, Hsia TC, Tsai KD, Shih CM, Hsu WH. Ultrasound in peripheral pulmonary air-fluid lesions. Color Doppler imaging as an aid in differentiating empyema and abscess. Chest. 2009 Jun;135(6):1426-1432. doi: 10.1378/chest.08-2188. Epub 2009 Mar 2. PMID 19255298